CLINICAL TRIAL: NCT00578331
Title: Safety Study of Olopatadine Nasal Spray
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C-05-69
Record Dates: First submitted 2007-12-19; First posted 2007-12-21 (Estimated); Results first posted 2010-02-03 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2010-02

CONDITIONS: Perennial Allergic Rhinitis
Keywords: rhinitis; perennial allergic rhinitis; allergic rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Perennial; Rhinitis; Rhinitis, Allergic | interventions — Olopatadine Hydrochloride; Nasal Sprays

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Olopatadine 0.6% Nasal Spray (Experimental): 2 sprays each nostril twice daily
  Interventions: Drug: Olopatadine 0.6% nasal spray
- Placebo Nasal Spray (Placebo Comparator): 2 sprays each nostril twice daily
  Interventions: Drug: Placebo Nasal Spray

INTERVENTIONS:
Drug: Olopatadine 0.6% nasal spray — 2 sprays each nostril twice daily
  Arms: Olopatadine 0.6% Nasal Spray
Drug: Placebo Nasal Spray — 2 sprays each nostril twice daily
  Arms: Placebo Nasal Spray

SUMMARY:
The purpose of this study is to determine whether olopatadine nasal spray is safe and effective when used for up to one year by patients with perennial allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed diagnosis of perennial allergic rhinitis who are 12 years and older

Exclusion Criteria:

* Age 11 years and younger

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 890 (Actual)
Dates: Start 2006-12; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Drake, Study Director — Alcon Research
Locations (1):
- Waco, Waco, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited between December 2006 and January 2007 at medical offices in the United States.
Pre-assignment Details: Patients were randomized at Visit 1 upon meeting inclusion/exclusion.
Period: Overall Study
Arm/Group | Placebo Nasal Spray | Olopatadine 0.6% Nasal Spray
Started | 445 | 445
Completed | 329 | 320
Not Completed | 116 | 125

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Nasal Spray | Olopatadine 0.6% Nasal Spray | Total
Number analyzed (Participants) | 445 | 445 | 890
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 53 | 46 | 99
  Between 18 and 65 years | 383 | 388 | 771
  >=65 years | 9 | 11 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 296 | 282 | 578
  Male | 149 | 163 | 312

OUTCOME MEASURES:

1. Primary Outcome: Mean Response at Day 30 to the Patient-rated Relief Assessment Questionnaire
Description: Mean Patient-Rated Relief Assessment at Day 30. The patient-rated relief assessment (PRRA) was a 4-point scale with 1=Complete Relief; 2=Moderate Relief; 3=Mild Relief; and 4=No Relief.
Time Frame: day 30
Population: 29 patients had missing mean patient-rated relief assessment data.
Measure: Mean (Standard Deviation); unit: Unit on PRRA scale
Arm/Group | Placebo Nasal Spray | Olopatadine 0.6% Nasal Spray
Number analyzed (Participants) | 430 | 431
Unit on PRRA scale | 2.7 (0.9) | 2.5 (0.9)

2. Secondary Outcome: Average Number of Days of Rescue Medication Taken
Time Frame: Month 1 through Month 12
Population: 12 patients had missing average use of rescue medication data.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo Nasal Spray | Olopatadine 0.6% Nasal Spray
Number analyzed (Participants) | 439 | 439
Days | 10.2 (22.4) | 11.8 (26.6)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Placebo Nasal Spray | Olopatadine 0.6% Nasal Spray
Serious Adverse Events (participants affected / at risk) | 15/445 | 15/445
Other Adverse Events (participants affected / at risk) | 319/445 | 309/445
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Nasal Spray (N=445) | Olopatadine 0.6% Nasal Spray (N=445)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Cholecystectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 3 (3)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Genital prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hip dysplasia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Hysterectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 3 (4) | 2 (2)
Intervertebral disc operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Joint surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Peripheral embolism (Vascular disorders) | 0 (0) | 1 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroidectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Nasal Spray (N=445) | Olopatadine 0.6% Nasal Spray (N=445)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 126 (212) | 111 (189)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 65 (148) | 46 (97)
Headache (Nervous system disorders) | 56 (110) | 57 (123)
Rhinitis (Infections and infestations) | 73 (108) | 87 (126)
Upper respiratory tract infection (Infections and infestations) | 75 (102) | 73 (97)
Nasopharyngitis (Infections and infestations) | 67 (90) | 72 (98)
Sinusitis (Infections and infestations) | 58 (72) | 66 (96)
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 38 (52) | 46 (62)
Seasonal allergy (Immune system disorders) | 29 (62) | 28 (44)
Injury (Injury, poisoning and procedural complications) | 49 (61) | 31 (34)
Asthma (Respiratory, thoracic and mediastinal disorders) | 24 (33) | 29 (36)
Sinus headache (Nervous system disorders) | 23 (42) | 15 (21)
Cough (Respiratory, thoracic and mediastinal disorders) | 23 (29) | 23 (32)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 26 (29) | 21 (24)
Bronchitis (Infections and infestations) | 19 (21) | 23 (25)
Dysgeusia (Nervous system disorders) | 3 (3) | 29 (30)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other